CLINICAL TRIAL: NCT00181883
Title: Open-Label Study of Quetiapine for Mania In Preschool Children 4 to 6 Years of Age With Bipolar and Bipolar Spectrum Disorder
Brief Title: Quetiapine for Mania In Preschool Children 4 to 6 Years of Age With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Janet Wozniak, MD, Assistant Professor of Psychiatry at Harvard Medical School and at Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-P-001509
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-03

CONDITIONS: Bipolar Disorder; Mania
Keywords: children; bipolar disorder; quetiapine; preschoolers
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quetiapine (Experimental): 2.5 - 5.0mg/kg PO BID quetiapine
  Other Names:
  Seroquel
  Interventions: Drug: quetiapine

INTERVENTIONS:
Drug: quetiapine — 2.5 - 5.0mg/kg PO BID quetiapine
  Other Names: Seroquel

SUMMARY:
This is an 8-week open-label study aimed at assessing the effectiveness and tolerability of Quetiapine, in the treatment of preschool children aged 4 to 6 years with bipolar and bipolar spectrum disorder. This is an exploratory, pilot study, seeking to determine whether Quetiapine is efficacious and well tolerated in the treatment of preschoolers with pediatric bipolar and bipolar spectrum disorder in this age group. The study results will be used to generate hypotheses for a larger randomized controlled clinical trial with explicit hypotheses and sufficient statistical power.

DETAILED DESCRIPTION:
Seroquel is a psychotropic agent that affects multiple neurotransmitter receptors in the brain: serotonin 5HT1A and 5HT2, dopamine D1 and D2, histamine H1 (IC50=30nM), and adrenergic receptors.

This is an 8-week open-label study aimed at assessing the effectiveness and tolerability of Quetiapine, in the treatment of preschool children aged 4 to 6 years with bipolar and bipolar spectrum disorder. This is an exploratory, pilot study, seeking to determine whether Quetiapine is efficacious and well tolerated in the treatment of preschoolers with pediatric bipolar and bipolar spectrum disorder in this age group. The study results will be used to generate hypotheses for a larger randomized controlled clinical trial with explicit hypotheses and sufficient statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 4-6 years of age.
* Subjects must have a DSM-IV diagnosis of bipolar I, bipolar II disorder or bipolar spectrum disorder and currently displaying manic, hypomanic, or mixed symptoms (with or without psychotic features) according to the DSM-IV based on clinical assessment and confirmed by structured diagnostic interview (Kidd Schedule of Affective Disorders and Schizophrenia Epidemiological Version). Bipolar spectrum disorder (or sub-threshold bipolar disorder) is operationalized as having severe mood disturbance, which meets DSM-IV Criteria A for bipolar disorder but meet fewer elements in criteria B (only require 2 items for elation category and 3 for irritability).
* Subjects and their legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Subjects and their legal representative must be considered reliable.
* Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document.
* Subjects must have an initial score on the Young Mania Rating Scale (Y-MRS) total score of at least 20.
* Subject must be able to participate in mandatory blood draws.
* Subjects with comorbid Attention Deficit Hyperactivity Disorder (ADHD), Oppositional Defiant Disorder (ODD), Conduct Disorder (CD), anxiety and depressive disorders will be allowed to participate in the study provided they do not meet for any of the exclusionary criteria.
* For concomitant stimulant therapy used to treat ADHD, subjects must have been on a stable dose of the medication for 1 month prior to study enrollment. The dose of the stimulant therapy will not change throughout the duration of the study.

Exclusion Criteria:

* Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
* Serious, unstable illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
* Uncorrected hypothyroidism or hyperthyroidism.
* History of severe allergies or multiple adverse drug reactions.
* Non-febrile seizures without a clear and resolved etiology.
* Leukopenia or history of leukopenia without a clear and resolved etiology.
* Judged clinically to be at serious suicidal risk.
* Any other concomitant medication with primarily central nervous system activity other than specified in Concomitant Medication portion of the protocol.
* A non-responder or a history of intolerance to an adequate trial of Quetiapine(2 months or more at an adequate dose) as determined by the clinician.
* Current diagnosis of schizophrenia.
* Non English speaking subjects will not be allowed into the study for the following reasons: a) the assessment instruments are not available and have not been adequately standardized in other languages; b) our clinical trials facility is located in Cambridge and not in the MGH main campus without the availability of translators; c) psychiatric questionnaires and evaluations are taxing and adding the complexity of a translator has the potential to make the patient experience even more exhausting.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wozniak, MD, Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Derived] Joshi G, Petty C, Wozniak J, Faraone SV, Doyle R, Georgiopoulos A, Hammerness P, Walls S, Glaeser B, Brethel K, Yorks D, Biederman J. A prospective open-label trial of quetiapine monotherapy in preschool and school age children with bipolar spectrum disorder. J Affect Disord. 2012 Feb;136(3):1143-53. doi: 10.1016/j.jad.2011.09.042. Epub 2011 Oct 28. PMID 22035648

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quetiapine
Started | 30
Completed | 20
Not Completed | 10
Not completed — Lack of Efficacy | 2
Not completed — Treatment Limiting AEs | 3
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Quetiapine
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 5.2 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Bipolar Symptoms as Measured by Reduction in Young-Mania Rating Scale (Y-MRS) Total Score
Description: The Y-MRS is used to evaluate mania symptoms in children and adolescents. Items on the scale are rated from 0-4 or 0-8, with higher values indicating greater severity. The minimum (least severe) total score is 0, with the maximum (most severe) score is 60.
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Quetiapine
Number analyzed (Participants) | 30
Units on a scale | -14.5 (11.4)

ADVERSE EVENTS:
Arm/Group | Quetiapine
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine (N=30)
suicidal ideation (Psychiatric disorders) | 1 (1) — 1 subject was terminated due to a serious adverse event possibly related to study medication. The subject had an increase in underlying symptoms of bipolar disorder, experiencing passive suicidal ideation (also present before participation).
OTHER ADVERSE EVENTS (reported when occurring in more than 3.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine (N=30)
chin/elbow abrasions (Injury, poisoning and procedural complications) | 1 (1)
injury (fall) (Injury, poisoning and procedural complications) | 1 (1)
agitation (General disorders) | 2 (2)
anxious/figety (General disorders) | 1 (1)
blurry vision (General disorders) | 1 (1)
cold symptoms (General disorders) | 2 (2)
congested (Respiratory, thoracic and mediastinal disorders) | 6 (8)
constipation (Gastrointestinal disorders) | 3 (6)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
daytime sleepiness (General disorders) | 3 (5)
depressed mood (General disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
enlarged gland, right side of neck (General disorders) | 1 (1)
enuresis (General disorders) | 4 (6)
epistasis (nose bleeding) (General disorders) | 1 (1)
fever (General disorders) | 2 (3)
flu (General disorders) | 1 (1)
headache (General disorders) | 4 (8)
increased appetite (General disorders) | 4 (11)
insect bite (General disorders) | 1 (1)
irritable (General disorders) | 1 (2)
lethargy (General disorders) | 2 (3)
minor burn on arm (General disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2)
pallor (General disorders) | 1 (1)
perseveration (General disorders) | 1 (1)
sedation (General disorders) | 2 (4)
skin irritation (Skin and subcutaneous tissue disorders) | 2 (2)
sleepiness (General disorders) | 8 (13)
slurred speech (General disorders) | 1 (3)
somnolence (General disorders) | 1 (1)
sore throat (General disorders) | 3 (5)
stomach ache (Gastrointestinal disorders) | 4 (6)
sunburn (Skin and subcutaneous tissue disorders) | 1 (1)
teary (General disorders) | 1 (2)
thirsty/dry mouth (General disorders) | 1 (1)
tiredness (General disorders) | 6 (11)
vomiting (Gastrointestinal disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No